CLINICAL TRIAL: NCT06452147
Title: Anesthesia and Perioperative Neurocognitive Disorders in the Elderly Patients Undergoing Hip Fracture Surgery Platform Trial (ANDES Platform Trial): A Pragmatic Multi-arm, Adaptive, Open Label, Multicenter Randomized Controlled Platform Trial to Assess the Effect of Different Enhance Anesthesia Technique in Perioperative Neurocognitive Function, as Compared to Standard Anesthesia Care in the Elderly Patients Undergoing Hip Fracture
Brief Title: Anesthesia and Perioperative Neurocognitive Disorders in the Elderly Patients Undergoing Hip Fracture Surgery Platform Trial (ANDES Platform Trial)
Acronym: ANDES platform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Zhejiang Provincial People's Hospital/ People's Hospital of Hangzhou Medical College (Unknown); The 1st Affiliated Hospital of Wenzhou Medical University (Unknown); Ningbo No.2 Hospital (Other); Ningbo No.6 Hospital (Other); Taizhou Hospital of Zhejiang Province affiliated to Wenzhou Medical University (Other); Taizhou Hospital (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Lishui Country People's Hospital (Other); The Fifth Hospital Affiliated to Wenzhou Medical University/ Lishui Central Hospital (Unknown); Jinhua Municipal Central Hospital (Other); Dongyang People's Hospital (Other); People's Hospital of Quzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2024-03-112
Record Dates: First submitted 2024-05-28; First posted 2024-06-11 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia; Hip Fractures; Dementia; Cognitive Impairment; Cognitive Decline
MeSH Terms: conditions — Hip Fractures; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nerve block + standard anesthesia protocol (Experimental): (described in detail in sub-trial protocol 1)
  Interventions: Other: Nerve block+standard anesthesia; Drug: Bupivacaine liposome; Device: Ultrasound-guided nerve block
- Intravenous infusion of lidocaine + standard anesthesia protocol (Experimental): (described in detail in sub-trial protocol 2)
  Interventions: Drug: Intravenous lidocaine+standard anesthesia
- Standard anesthesia protocol (No Intervention): (If an intervention was found to be effective in the interim analysis, the executive committee will decide whether to add it to the standard anesthesia protocol.)

INTERVENTIONS:
Other: Nerve block+standard anesthesia — 1. Receive nerve block as soon as possible after randomization;
  2. Ultrasound-guided nerve block is recommended, with the iliacfascia block recommended as the blocking site;
  3. It is recommended to use 1.33% bupivacaine liposome (long-acting), and the maximum dose should not exceed 133mg; or regular local anesthetic (bupivacaine or ropivacaine, etc.) with electronic analgesic pumping infusion; or multiple single injections of regular local anesthetics should be used to maintain the continuity of nerve block effect.
  Arms: Nerve block + standard anesthesia protocol
Drug: Intravenous lidocaine+standard anesthesia — 1. Subjects randomly assigned to Lidocaine Group (Group L) will be given ECG monitoring, oxygen saturation monitoring, blood pressure monitoring and an open intravenous route on the morning of the surgery. It is recommended to start the infusion of Lidocaine as soon as possible in the ward.
  2. It is recommended to use portable electronic infusion pump for drug delivery. The loading dose is 1mg/kg, and the maintenance dose range is 1~2mg/kg/h. The specific dosage is determined by the anesthesiologist based on the patient's condition. The infusion ends when the patient leaves the Post-anesthesia care unit after surgery, and the infusion time and total amount should be recorded.
  Arms: Intravenous infusion of lidocaine + standard anesthesia protocol
Drug: Bupivacaine liposome — 1.33% bupivacaine liposome
  Arms: Nerve block + standard anesthesia protocol
Device: Ultrasound-guided nerve block — Ultrasound-guided nerve block
  Arms: Nerve block + standard anesthesia protocol

SUMMARY:
Anesthesia and perioperative Neurocognitive Disorders in the Elderly patients undergoing hip fracture Surgery platform trial (ANDES platform trial): A pragmatic multi-arm, adaptive, open label, multicenter randomized controlled platform trial to assess the effect of different enhance anesthesia technique in perioperative neurocognitive function, as compared to standard anesthesia care in the elderly patients undergoing hip fracture

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 years and older.
2. Patients with unilateral hip fracture (including femoral neck, femoral head, intertrochanteric and subtrochanteric fractures) are scheduled for surgical treatment.
3. American Society of Anesthesiologists (ASA) physical status IV or below.
4. The patients or family members provide written informed consent.
5. Additional inclusion criteria may pertain to specific interventions and will be described in relevant sub-protocols.

Exclusion Criteria:

1. Patients with multiple trauma or fractures (excluding trauma that the researcher judges will not affect the patient's overall recovery, such as simple spinal compression fractures, mild soft tissue contusions, fractures of hands and feet, etc.);
2. Two or more anesthetic surgeries are required.
3. Petients with an obvious history of head trauma (such as loss of consciousness for more than 5 minutes, post-traumatic amnesia, etc.);
4. Patients who the researcher believes are unable to complete the assessment of primary outcome;
5. Additional exclusion criteria may pertain to specific interventions and will be described in relevant sub-protocols.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1860 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Neurocognitive Disorders (NCD) events rate during the first 7 postoperative days | during the first 7 postoperative days
  Neurocognitive Disorders includes:
  1. Postoperative delirium (POD) was mesaured by 3D-CAM;
  2. Neurocognitive decline was mesaured within 7 postoperative days by: Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA), and neuropsychological tests containing 5 cognitive latitudes (1. digit span test (DST); 2. trail making test (TMT); 3. Boston naming test (BNT); 4. auditory verbal learning test-Huashan version (AVLT-H)；5. clock drawing test (CDT).）, and active report of patients or family members).

SECONDARY OUTCOMES:
Subtypes, severity, and duration of delirium | during the first 7 postoperative days
  Using CAM-S, and in units of days from the onset of delirium symptoms to the disappearance of symptoms or when the patient is discharged.
Neurocognitive decline in postoperative 7 days | during the first 7 postoperative days
  Neurocognitive decline was mesaured by: Mini-Mental State Examination (MMSE) or Montreal Cognitive Assessment (MoCA), or neuropsychological tests containing 5 cognitive latitudes (1. digit span test (DST); 2. trail making test (TMT); 3. Boston naming test (BNT); 4. auditory verbal learning test-Huashan version (AVLT-H)；5. clock drawing test (CDT).）, or active report of patients or family members.
Delayed neurocognitive recovery during 30 postoperative days | during 30 postoperative days
  This was mesaured by: Mini-Mental State Examination (MMSE) or Montreal Cognitive Assessment (MoCA), or neuropsychological tests containing 5 cognitive latitudes (1. digit span test (DST); 2. trail making test (TMT); 3. Boston naming test (BNT); 4. auditory verbal learning test-Huashan version (AVLT-H)；5. clock drawing test (CDT).）, or active report of patients or family members.
Hospital Anxiety and Depression Scale (HADs) | during postoperative one year
Acute pain before surgery | 1, 2, 3 days after surgery
  Using Visual Analogue Scale (VAS)
Length of hospitalization | days from admission to discharge, an average of 7 days
Complications (except cognitive impairment) | during postoperation 30 days
  including pulmonary infection, myocardial infarction, renal failure, gastrointestinal obstruction, etc.
Mortality | 30 days
Days at home up to 30 days after surgery (DAH30) | up to 30 days after surgery
Score of EuroQol Five Dimensions Questionnaire (EQ-5D) | 1 week before fracture (review); 1 month; 6 months; and 12 months after surgery.
  using EQ-5D to measure quality of life
Incidence of postoperative Neurocognitive Disorders (NCD) | within 1 year after surgery (long-term)
  This was mesaured within 7 postoperative days by: Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA), and neuropsychological tests containing 5 cognitive latitudes (1. digit span test (DST); 2. trail making test (TMT); 3. Boston naming test (BNT); 4. auditory verbal learning test-Huashan version (AVLT-H)；5. clock drawing test (CDT).), and active report of patients or family members).
Severity of postoperative Neurocognitive Disorders (NCD) | within 1 year after surgery (long-term)
  Includes major and mild postoperative NCD
Type of postoperative Neurocognitive Disorders (NCD) | within 1 year after surgery (long-term)
  Using Hachinski Ischemic Scale (HIS) combined with clinical symptoms and auxiliary examination to mesaure the type of postoperative NCD. HIS ≥7 was considered as vascular cognitive impairment.
Instrumental Daily Living Ability Scale (IADL) | within 1 year after surgery (long-term)
  IADL ≤6 is normal
1-year all-cause mortality | 1-year after surgery
Economic indicators | during the entire trial, an average of 1 year.
  * Hospitalization fees;
  * Preoperative fees;
  * Anesthesia fees;
  * Surgery fees;
  * Post-operative fees;
  * Post-discharge medical expenses.

OTHER OUTCOMES:
Incidence of adverse events | during hospitalization, an average of 7 days; through entire trial, an average of 1 year.
  We will collect the following known potential risks of general and local anesthesia from the start of the intervention to the subject's discharge and assess the overall incidence:
  1. cardiopulmonary resuscitation;
  2. Malignant hyperthermia or anaphylaxis;
  3. Aspiration pneumonia ;
  4. Epidural hematoma ;
  6) Patients who did not need mechanical ventilation before surgery continued with unplanned mechanical ventilation for more than 6 hours after surgery; 7) Other adverse events during postoperative hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affilliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No